CLINICAL TRIAL: NCT02527070
Title: Evaluating an Optical Index (Minimum Rise Time) as a Measure for the State of Microvessels
Brief Title: Evaluating the State of Microvessels by Minimum Rise Time (MRT01)
Acronym: MRT01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Afeka, The Tel-Aviv Academic College of Engineering (Other)
Collaborators: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2080-15-SMC
Record Dates: First submitted 2015-07-28; First posted 2015-08-18 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Red LED (Experimental): Light emitting diodes, 670 nm, 50 mW/cm2, Quantum Warp10 (Quantum Devices Inc, Barneveld, WI, USA); RESPeRATE; Heat/cold provocation
  Interventions: Device: RESPeRATE (Paced Breathing); Device: Quantum Warp10 (Red LED); Other: Heat/cold provocation
- Near Infrared LED (Active Comparator): Light emitting diodes, 830 nm, 55 mW/cm2, Omnilux new-U (Photomedex, Horsham, PA, USA); RESPeRATE; Heat/cold provocation
  Interventions: Device: RESPeRATE (Paced Breathing); Device: Omnilux new-U (Near Infrared LED); Other: Heat/cold provocation

INTERVENTIONS:
Device: RESPeRATE (Paced Breathing) — The subjects will be guided by a digital metronome to breath at 15, 10, and 6 breaths/min for 2 minutes each using the metronome function of the device RESPeRATE (InterCure, Israel) that guides breathing using musical tones played at selectable rhythm.
Device: Quantum Warp10 (Red LED)
  Arms: Red LED
Device: Omnilux new-U (Near Infrared LED)
  Arms: Near Infrared LED
Other: Heat/cold provocation — Immersion of one foot in a warm water bath ( 43-45 degrees C) for few seconds and then immersion of the same foot in cold water bath (5-7 degrees C) for 1 min.

SUMMARY:
Photoplethysmography (PPG) is a simple uncalibrated optical method of monitoring variations in skin blood volume. The objective of the current study is to investigate a potential relationship between MRT (minimum rise time, in time units) a measure derived from PPG and the state of microvessels.

This study includes a 1-2 hour single session per subject during which PPG and other microvascular and systemic variables will be monitored in response to non-invasive interventions that are known to elicit microvascular responses.

DETAILED DESCRIPTION:
Photoplethysmography (PPG) is a simple uncalibrated optical method of monitoring variations in skin blood volume. A major limitation of PPG is the lack of a quantitative method for calibrating this signal. A method that provides an absolute measure (in time units) called 'minimum rise time' (MRT) was published in 1985 by Dr. Benjamin Gavish, one of the study investigators. However, a possible relationship between MRT and the state of arterioles that determines the microvascular flow has never been investigated. Such relationship, if validated, could have clinical impact in noninvasive diagnosis of vascular diseases and monitoring microvascular response to treatments that affect at both clinic and home setting.

The objective of the current study is to investigate a potential relationship between variations of MRT (minimum rise time, in time units) and microcirculatory variables induced by interventions that are expected to have acute effect on the state of arterioles and the tissue oxygenation.

This study includes a single 1-2 hour session per subject, during which PPG and other microvascular and systemic variables will be monitored in healthy volunteers in response to a number of non-invasive interventions/device that are approved for clinical use and known to elicit microvascular responses. These interventions are applied consecutively, include breathing at different rates, low power visible light in the red-to-near-infrared range, and local temperature changes. The experimental sessions will be conducted at the Afeka College by the study investigators.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females, between 18 and 65 years of age.
2. Willing to sign informed consent.

Exclusion Criteria:

1. Currently smoking
2. Any abnormal skin condition in the area of light irradiation.
3. Pregnant having given birth less than 3 months ago, and/or breastfeeding.
4. Having a history of diseases stimulated by heat, such as recurrent Herpes Simplex in the treated area, unless treatment is conducted following a prophylactic regimen.
5. Having any illness that might affect the vasculature, such as diabetes (type I or II)
6. Suffering from significant concurrent illness, such as cardiac disorders, , or pertinent neurological disorders.
7. As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2015-09; Primary Completion 2016-06 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
MRT as measured from finger Photoplethysmography in response to changes in breathing rate | Change from baseline to up to 1 minute after termination of 2 minutes of constant breathing rate (15, 10, and 6 breath/min)
MRT as measured from finger Photoplethysmography in response to light source | Change from immediately before exposure to light source to up to 10 minutes after exposure to light source
MRT as measured from finger Photoplethysmography in response to temperature changes | Change from immediately before exposure to temperature provocations to up to 2 minutes after exposure to warm water, and up to 2 minutes after exposure to cold water

SECONDARY OUTCOMES:
Capillary blood flow (red blood cell velocity or flux in 'perfusion units') as measured by laser doppler | At baseline, 1 minute after each changes in breathing rate, 5 and 10 minutes after exposure to light source, 1 minutes after each exposure to temperature changes
Transcutaneous oxygen pressure (tcpO2 in mmHg) | At baseline, 1 minute after each changes in breathing rate, 5 and 10 minutes after exposure to light source, 1 minutes after each exposure to temperature changes

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Halak, MD, Principal Investigator — Sheba Medical Center; Zehava Blechman, PhD, Study Director — Afeka, Tel-Aviv Academic College of Engineering
Locations (1):
- Afeka, Tel-Aviv Academic College of Engineering, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Gavish B. Plethysmographic characterization of vascular wall by a new parameter--minimum rise-time: age dependence in health. Microcirc Endothelium Lymphatics. 1986-1987;3(3-4):281-96. PMID 3431526